CLINICAL TRIAL: NCT03712254
Title: Phenytoin as Treatment for Acute Exacerbations of Trigeminal Neuralgia - a Prospective Systematic Study of 30 Patients
Brief Title: Phenytoin as Treatment for Acute Exacerbations of Trigeminal Neuralgia - a Prospective Systematic Study of 20 Patients
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Lars Bendtsen, Associate professor, Danish Headache Center
Other Study IDs: H-18023737
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Trigeminal Neuralgia
Keywords: acute pain, fosphenytoin
MeSH Terms: conditions — Trigeminal Neuralgia; Acute Pain | interventions — fosphenytoin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Fosphenytoin — Patients with trigeminal neuralgia that due to acute exacerbations of trigeminal neuralgia pain are admitted for fosphenytoin loading are the subjects of interest.

SUMMARY:
The nature of trigeminal neuralgia (TN) is fluctuating and patients can experience periods of complete remission of pain as well as periods with excessive pain. TN is often triggered by innocuous intra- and extraoral stimuli such as chewing. Since the first-line prophylactic drugs, i.e. carbamazepine and oxcarbazepine, are administered orally, medical treatment of TN can be problematic in periods of exacerbation. In cases of severe exacerbation, patients oftentimes become dehydrated and anorectic as eating and drinking will evoke pain. Treatment with drugs administered intravenously is needed in such situations. Phenytoin was the first drug to be used for TN but it is rarely used as long-time preventative because of frequent side-effects associated with long-term use. However, phenytoin has the advantage over other drugs, that it can be administered also intravenously as fosphenytoin (the prodrug of phenytoin).

By clinical experience the efficacy is very good. However, evidence of the treatment is lacking as only case reports including a total of 5 patients described the effects and side effects with pain relief lasting two days. By providing solid observational evidence, the treatment can be considered for incorporation in local and international treatment guidelines.

The aim of the study is to test the hypothesis that fosphenytoin loading reduces TN pain with at least 50 % in 80% of patients with trigeminal neuralgia experiencing exacerbation of TN pain.

The study is a descriptive prospective observational pilot study with 3 months followup period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Must be able to give signed informed consent prior to study entry.
* Must fulfill the ICHD-3 diagnostic criteria for TN. Both patients with purely paroxysmal TN and patients with TN with concomitant persistent facial pain will be included.
* MRI of the brain, brainstem and trigeminal nerve or patient is willing to undergo MRI in the days and weeks following admission.
* Must be able to adhere to the study protocol and understand either Danish or English.

Exclusion Criteria:

* Psychiatric or mental illness or condition that might interfere with the ability of the patients to fill in the Informed Consent.
* Contraindications for phosphenytoin loading such as sick sinus syndrome, atrioventricular block and hepatic insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with trigeminal neuralgia admitted for fosphenytoin loading due to acute exacerbations of trigeminal neuralgia pain.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Degree of acute pain relief | Primary outcome is measured app. 24 hours after fosphenytoin loading.
  Degree of pain relief measured by the verbal numeric rating scale of pain 24 hours after treatment compared with 24 hours before treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Rigshospitalet - Glostrup, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Andersen ASS, Heinskou TB, Asghar MS, Rossen B, Noory N, Smilkov EA, Bendtsen L, Maarbjerg S. Intravenous fosphenytoin as treatment for acute exacerbation of trigeminal neuralgia: A prospective systematic study of 15 patients. Cephalalgia. 2022 Oct;42(11-12):1138-1147. doi: 10.1177/03331024221094536. Epub 2022 Apr 25. PMID 35469443